CLINICAL TRIAL: NCT06673862
Title: Changes in Pulse-Oximetry Perfusion Index Induced by Tidal Volume Challenge Versus Fluid Volume Challenge to Detect Preload Responsiveness in Mechanically Ventilated Patients With Low Tidal Volume: A Prospective Observational Study
Brief Title: Changes in Pulse-Oximetry Perfusion Index Induced by Tidal Volume Challenge Versus Fluid Volume Challenge to Detect Preload Responsiveness in Mechanically Ventilated Patients With Low Tidal Volume
Status: Enrolling by invitation | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Salwa Abbas Awad Eltahawy, Assistant Lecturer of Critical Care Medicine, Benha University
Other Study IDs: MD 2-8-2024
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: To Assess the Ability of PI to Detect Preload Responsiveness
Keywords: fluid responsiveness; VTI; PI; tidal volume challenge; fluid challenge; perfusion index; velocity time index; preload responsiveness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary goal of this study was to assess the ability of PI changes induced by a Vt challenge or fluid challenge test to detect preload responsiveness in critically ill adult patients on mechanical ventilation with low-tidal volume.

The secondary aims were (i) to compare the changes in PI with VTI during a Vt challenge test (ii) to compare the changes in VTI and PI during a volume expansion challenge test, (iii) to compare the Vt-induced changes in PI to changes induced by fluid challenge test, (iv) to compare the Vt-induced changes in VTI to changes induced by fluid challenge test.

ELIGIBILITY:
Inclusion Criteria:

Patients of both genders aged 18 years or older Invasive mechanical ventilation in assist controlled mode with a Vt of 6 mL/kg PBW, Patients with circulatory failure Decision by the clinicians in charge to assess preload responsiveness through a Vt Challenge and a Fluid Challenge test.

Patients in sinus rhythm

Exclusion Criteria:

Open chest Pulmonary hypertension Poor lung compliance (Crs <30 ml/cmH2O) Obesity (BMI≥35) Pregnancy Intraabdominal hypertension Prone position Atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted on 75 mechanically ventilated patients with circulatory failure.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The ability of perfusion index to detect preload responsiveness | Approximately one hour
  The primary goal of this study was to assess the ability of PI changes induced by a Vt challenge or fluid challenge test to detect preload responsiveness in critically ill adult patients on mechanical ventilation with low-tidal volume.

SECONDARY OUTCOMES:
Compare the changes in PI with VTI during a Vt challenge test | Approximately one hour
Compare the changes in VTI and PI during a volume expansion challenge test | Approximately one hour
Compare the Vt-induced changes in PI to changes induced by fluid challenge test | Approximately one hour

OTHER OUTCOMES:
Compare the Vt-induced changes in VTI to changes induced by fluid challenge test | Approximately one hour

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mostafa Abdelhamid, Principal Investigator — Benha University; Samar Rafik Mohamed Amin, Principal Investigator — Benha University; Mona Sobhy Emara, Principal Investigator — Benha University; Salwa Abbas Awad Eltahawy, Principal Investigator — Benha University
Locations (1):
- Faculty of Medicine- Benha University, Banhā, Al-Qalyubia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT06673862/Prot_SAP_000.pdf